CLINICAL TRIAL: NCT00234949
Title: A Comparative Study of the Safety, Tolerability, and Efficacy of Cefdinir and Cephalexin for the Treatment of Subjects With Mild to Moderate Uncomplicated Skin and Skin Structure Infections
Brief Title: A Study to Compare Cefdinir and Cephalexin for the Treatment of Mild to Moderate Uncomplicated Skin Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M04-699
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Mild to Moderate Uncomplicated Skin and Skin Structure Infections
Keywords: Cefdinir; Cephalexin; Skin Infection
MeSH Terms: conditions — Cellulitis | interventions — Cefdinir; Cephalexin

INTERVENTIONS:
Drug: cefdinir
Drug: cephalexin

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of cefdinir to that of cephalexin in patients with mild to moderate uncomplicated skin/skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female subjects > 13 years old.
* A female subject must be non-lactating and at no risk for pregnancy.
* Diagnosis of USSSI with 2 or more of the following local signs and symptoms:

  * Pain/tenderness
  * Swelling
  * Erythema
  * Localized warmth
  * Purulent drainage/discharge
  * Induration
  * Regional lymph node swelling or tenderness
  * Extension of redness
* Acceptable USSSI include, but are not limited to:

  * Cellulitis
  * Erysipelas
  * Impetigo
  * Simple abscess
  * Wound infection
  * Furunculosis
  * Folliculitis
* A sample for microbiologic culture must be obtained from the primary infection site within 48 hours prior to study drug administration.

Exclusion Criteria

* Medical history of hypersensitivity or allergic reaction to penicillin and/or cephalosporin (including cefdinir and cephalexin) antibiotics according to the judgment of the Investigator.
* Subject with a complicated skin and skin structure infection as judged by the investigator.
* A chronic or underlying skin condition at the site of infection (e.g., a secondary infected atopic dermatitis or eczema) or infections involving prosthetic materials (e.g., catheter tunnel infections, orthopedic hardware).
* A wound secondary to burn injury or acne vulgaris.
* Any infection site that requires:

  * intraoperative surgical debridement;
  * excision of infected lesions or body parts.
* Infections that can be treated by surgical incision alone according to the judgment of the Investigator.
* Any other infection that necessitates the use of additional concomitant oral or parenteral antibiotic therapy.
* Known significant renal or hepatic impairment indicated by:

  * Serum Creatinine > 2.0 mg/dL (176.8 mol/L)
  * SGOT (AST) > 3x the upper limit of the reference range
  * SGPT (ALT) > 3x the upper limit of the reference range
  * Alkaline Phosphatase > 2x the upper limit of the reference range
  * Total Bilirubin > 2x the upper limit of the reference range
* Underlying condition and/or disease that, according to the judgment of the Investigator, would be likely to interfere with completion of the course of study drug therapy or follow-up.
* The Investigator considers the subject an unsuitable candidate for cefdinir or cephalexin administration

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380
Dates: Start 2005-03

PRIMARY OUTCOMES:
Clinical cure rate

SECONDARY OUTCOMES:
Adverse event rates
Bacteriologic cure rates
Patient reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott